CLINICAL TRIAL: NCT07022847
Title: The Value of Pleth Variability Index in Predicting Hypotension During Maintenance Hemodialysis: A Prospective Observational Multicenter Study
Brief Title: Pleth Variability Index for Predicting Low Blood Pressure During Maintenance Hemodialysis
Acronym: PVI-HD
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Wannan Medical College (Other)
Collaborators: Wuhu City Second People's Hospital (Other); Wuhu County Traditional Chinese Medicine Hospital (Other)
Responsible Party: Principal Investigator, Qiancheng Xu, Principal Investigator, First Affiliated Hospital of Wannan Medical College
Other Study IDs: 2025-61
Record Dates: First submitted 2025-06-07; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Hypotension and Shock; Hemodialysis; End-Stage Renal Disease Requiring Haemodialysis; Intradialytic Hypotension
Keywords: Pleth Variability Index; Hemodialysis; Intradialytic Hypotension; Blood Pressure Monitoring; End-Stage Renal Disease; Non-invasive Monitoring; Predictive Marker; Maintenance Dialysis
MeSH Terms: conditions — Hypotension; Shock; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Maintenance Hemodialysis Patients: Adult patients aged 18 to 80 years who have been receiving maintenance hemodialysis for more than 3 months. All participants will be monitored for blood pressure and Pleth Variability Index (PVI) measurements before and during hemodialysis sessions. The occurrence of intradialytic hypotension and its association with PVI will be evaluated.
  Interventions: Other: Non-invasive Monitoring

INTERVENTIONS:
Other: Non-invasive Monitoring — All participants will undergo non-invasive measurement of Pleth Variability Index (PVI) and routine blood pressure monitoring before and during hemodialysis sessions. No treatment or experimental intervention will be applied.

SUMMARY:
What is this study about? We are studying whether the Pleth Variability Index (PVI)-a simple, non-invasive measurement from a pulse oximeter-can help predict low blood pressure (hypotension) during routine maintenance hemodialysis. Low blood pressure during dialysis is a common and potentially serious complication. Our goal is to find out if monitoring PVI can help identify patients at risk, so that early action can be taken.

Who can join? Adults aged 18 to 80 years. Patients who have been receiving maintenance hemodialysis regularly for more than 3 months.

Those who are willing and able to participate and sign an informed consent form.

Who cannot join? Patients with severe heart rhythm problems, severe peripheral circulation problems, or swelling that makes PVI measurement unreliable.

Patients who are pregnant or breastfeeding. Patients allergic to the dialysis filter or unable to cooperate with the study procedures.

What will happen during the study? PVI Measurement: Your PVI will be checked with a simple fingertip device before starting dialysis and again 30 minutes after dialysis begins.

Blood Pressure Monitoring: Your blood pressure will be closely watched throughout the dialysis session.

Data Collection: Information about your age, medical history, medications, lab results, dialysis settings, and other standard measurements will be recorded.

What are the benefits and risks? Benefits: By identifying patients at higher risk for low blood pressure during dialysis, the study may lead to safer and more comfortable dialysis treatment in the future.

Risks: All measurements used in this study are safe and non-invasive, with no extra risk compared to routine care.

Your Rights and Safety Participation is completely voluntary-you may leave the study at any time without affecting your medical care.

The study has been reviewed and approved by the hospital's ethics committee. Your privacy and personal data will be strictly protected.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 80 years.
* Diagnosis of end-stage renal disease and undergoing maintenance hemodialysis for more than 3 months.
* Able and willing to provide informed consent and comply with study procedures.

Exclusion Criteria:

* Severe cardiac arrhythmias or significant peripheral vascular disease that may interfere with PVI measurements.
* Local edema, skin lesions, or other conditions that prevent accurate PVI monitoring.
* History of hemodynamic instability unrelated to dialysis.
* Pregnant or breastfeeding women.
* Known allergy or contraindication to materials used in the hemodialysis circuit.
* Unable to cooperate with study procedures.
* Participation in another interventional clinical study within the past 30 days.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 to 80 years with end-stage renal disease who have been receiving maintenance hemodialysis for more than three months at participating dialysis centers. Participants are required to be able to provide informed consent and cooperate with study procedures.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Predictive Value of PVI for Intradialytic Hypotension | Pre-dialysis (baseline), and 60 minutes after the start of a single hemodialysis session (total duration up to 4 hours).
  PVI measured at baseline (pre-dialysis) and at 60 minutes after the start of hemodialysis.
  The sensitivity, specificity, and area under the receiver operating characteristic (ROC) curve of PVI measured before and during hemodialysis in predicting hypotension events.
Predictive Value of Percentage Change in Pleth Variability Index (%PVi) for Intradialytic Hypotension | From pre-dialysis (baseline) to 60 minutes after the start of a single hemodialysis session (total duration up to 4 hours).
  The ability of the percentage change in PVI (%PVi) between pre-dialysis and 60minutes after the start of dialysis to predict intradialytic hypotension. This will be evaluated using sensitivity, specificity, and area under the ROC curve analysis.

SECONDARY OUTCOMES:
Incidence of Intradialytic Hypotension | Up to 1 dialysis session (4 hours)
  The proportion of hemodialysis treatments in which patients develop hypotension, defined as a decrease in systolic blood pressure of ≥20 mmHg
Predictive Value of Change in Pleth Variability Index (dPVi) for Intradialytic Hypotension | From pre-dialysis (baseline) to 60 minutes after the start of a single hemodialysis session (total duration up to 4 hours).
  The ability of the absolute difference in PVI (dPVi) between pre-dialysis and 60minutes after the start of dialysis to predict intradialytic hypotension. This will be evaluated using sensitivity, specificity, and area under the ROC curve analysis.
Correlation Between PVI, dPVi, %PVi and Changes in Blood Pressure | Pre-dialysis (baseline) and 60 minutes after the start of a single hemodialysis session (total duration up to 4 hours).
  Assessment of the statistical correlation between PVI parameters (PVI, dPVi, and %PVi) and changes in blood pressure, including systolic blood pressure, diastolic blood pressure, and mean arterial pressure, during the dialysis session. Blood pressure changes will be calculated as the difference between pre-dialysis (baseline) and corresponding post-initiation time points (60 minutes). Correlation analyses will use Pearson or Spearman methods as appropriate.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Wannan Medical College (Yijishan Hospital of Wannan Medical College), Wuhu, Anhui, China

IPD SHARING:
Plan to Share IPD: No